CLINICAL TRIAL: NCT05999409
Title: Evaluation of the Effectiveness of Simulation Use in the Management of Normal Labor
Brief Title: Normal Birth Management and Use of Simulation
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Ondokuz Mayıs University (Other)
Collaborators: Tokat Gaziosmanpasa University (Other)
Responsible Party: Principal Investigator, Serap Ozturk Altinayak, assistant professor, Ondokuz Mayıs University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: 22-KAEK-166
Record Dates: First submitted 2023-08-02; First posted 2023-08-21 (Actual); Last update posted 2023-11-29 (Actual); Status verified 2023-11

CONDITIONS: Obstetric

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- d1 (Experimental): NBSAF's first rating on a full-reality birth simulator. During the first normal delivery practice of the student in the hospital environment, the second evaluation of NBSAF and the second application of SSSCSL and ESSBL were made.
  Interventions: Other: practice on birth simulator
- d2 (Experimental): An initial evaluation of NBSAF was performed on a medium reality labor stimulator. During the first normal delivery practice of the student in the hospital environment, the second evaluation of NBSAF and the second application of SSSCSL and ESSBL were made.
  Interventions: Other: practice on birth simulator
- d3 (control) (No Intervention): Without any simulation application, the second evaluation of NBSAF and the second application of SSSCSL and ESSBL were performed during the first normal delivery practice of the student in the hospital environment.

INTERVENTIONS:
Other: practice on birth simulator — making attempts at labor
  Other Names: d2=medium reality birth simulator
  Arms: d1; d2

SUMMARY:
The research; It is planned to evaluate the effectiveness of the use of simulation in the management of normal labor.

The research was designed in a quasi-experimental randomized controlled type. The research is carried out in the Department of Midwifery, Faculty of Health Sciences, in the 2022-2023 academic year. The sample of the study consists of all third-year students who enrolled in the Normal Birth and Postpartum Term course in the midwifery department for the first time (102 students who successfully passed the Prenatal I course in the 2021-2022 academic year. These students are in the next 2022-2023 academic year. Registered for the Post Term Course). In the literature; In experimental studies, it has been reported that a sample size of at least 30 people is required in order to perform parametric tests (24). In this study, the number of students in the groups was determined as 32, considering that they may have lost. Students were divided into three groups as experimental (d1= High Reality simulator), (d2= Medium Reality simulator) group and control group (d3= slide and video presentation). The study is carried out with 96 students in total. The students who met the inclusion criteria were given a sequence number and then randomly divided into 3 groups using the https://www.randomizer.org online randomization program.

Data collection tools: In data collection; Introductory Information Form (IIF), Normal Birth Skills Assessment Form (NBSAF), Student Satisfaction and Self-Confidence Scale in Learning (SSSCSL) and Evaluation of Simulation-Based Learning Scale (ESSBL) will be used.

DETAILED DESCRIPTION:
Introductory Information Form (IIF); It was created by the researchers by scanning the literature (11,25-28). This form includes the socio-demographic characteristics of the students, the presence of a health worker in the family, their normal birth practice status and their simulation training (age, graduated high school, monthly income, presence of a health worker in the family, normal birth practice monitoring and performance, simulation training). receiving status etc.) consists of a total of 10 questions.

Normal Birth Skill Assessment Form (NBSAF) It was created by the researchers by scanning the literature (29-31). In the form, there are 50 items about the steps that the student should do during the normal labor practice. Evaluation of the form is as "he did" and "did not" in relation to the student's implementation of the activities to be observed during the normal labor process steps. In the form, the student was given 2 points for each activity he did, while 0 points were given for the activities he did not do. The lowest score that can be obtained from the form is 0, and the highest score is 100. A high score will indicate high skill, and a low score will indicate low skill.

For the content validity of the NBSAF items, the opinions of 5 experts (2,3,32-34) who have researched on learning techniques related to the management of normal labor were consulted. The Lawshe technique was used to evaluate the content validity of the items in the form. According to the Lawshe technique, the minimum fit criterion was 0.99 for five experts (35). No item with a content validity ratio below 0.99 was detected. In order to test the intelligibility of the items, a pilot study was conducted with 10 students from another class who had no knowledge of the content, and the form was given its final form.

Student Satisfaction and Self-Confidence Scale in Learning (SSSCSL) The original scale was developed as 13 items by Jeffries and Rizzolo (2006), and the total number of items decreased to 12 during its adaptation to Turkish. The adaptation of the scale to Turkish was done by Ünver et al. (2017). The scale is a 5-point Likert type and consists of the sub-headings of "Satisfaction with Current Learning" and "Self-Confidence in Learning". The sub-title of satisfaction with current learning consists of 5 items, the sub-title of self-confidence in learning consists of 7 items and there is no negative item. The cronbach alpha value of the scale for "Satisfaction with Current Learning" is .85, while it is .77 for "Self-Confidence in Learning", it is .89 for the total scale. Scale scores; It is obtained by dividing the sum of the sub-dimensions by the number of items. As the total score obtained from the scale increases, student satisfaction and self-confidence in learning also increase.

Evaluation Scale of Simulation-Based Learning (ESSBL) The original scale was developed by Hung et al. (2016), and its Turkish validity and reliability were performed by Uslu and Yavuz van Giersbergen (2020). The Turkish validity and reliability of the scale consists of 5 sub-dimensions and 37 items. Responses are scored on a five-point Likert system, ranging from 1 (strongly disagree) to 5 (strongly agree), and the total score varies between 37-185. All statements in the scale are positive and there is no reverse coded item. Within the scope of the scale, the basic competencies that midwives and nurses should have; care process, patient safety, professional knowledge, communication and reflected behavior concepts are evaluated. An increase in the score obtained from the sub-dimensions in the scale means that the sub-dimension goal has been achieved for the student in the scenario (37).

ELIGIBILITY:
Inclusion Criteria:

* The research includes all third-year students who registered for the first time to the Normal Birth and Postpartum Term course in the midwifery department in the 2022-2023 academic year in the Department of Midwifery at the Faculty of Health Sciences.

Exclusion Criteria:

* Having any of the above criteria

Ages: 18 Years to 28 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 90 (Estimated)
Dates: Start 2022-10-10 (Actual); Primary Completion 2023-07-20 (Actual); Study Completion 2023-12-10 (Estimated)

PRIMARY OUTCOMES:
providing access to the number | through study completion, an average of 9 month
  enough practice by students

CONTACTS AND LOCATIONS:
Locations (1):
- Health Research and Training Hospital of Tokat Gaziosmanpaşa University, Tokat Province, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided
Data can be shared if requested from researchers.